CLINICAL TRIAL: NCT03504449
Title: Surgery Without Neoadjuvant Chemoradiotherapy Compared With Neoadjuvant Chemoradiotherapy for Rectal Cancer With Negative Circumferential Resection Margin Based on MRI Assessment, a Perspective Multicenter Randomized Controlled Trial
Acronym: SCRM-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Chairman of General Surgery, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRM-01
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Circumferential Resection Margin; Intraoperative Perforation of Rectum; Local Recurrence of Malignant Tumor of Rectum; Disease-free Survival; Overal Survival
MeSH Terms: interventions — Neoadjuvant Therapy

ARMS (2):
- surgery without neoadjuvant chemoradiotherapy (Experimental): For T3N1-2M0 rectal cancer with negative circumferential resection margin based on MRI assessment, recieve surgery without neoadjuvant chemoradiotherapy.
  Interventions: Other: neoadjuvant chemoradiotherapy
- surgery with neoadjuvant chemoradiotherapy (Experimental): For T3N1-2M0 rectal cancer with negative circumferential resection margin based on MRI assessment, recieve surgery following neoadjuvant chemoradiotherapy.
  Interventions: Other: neoadjuvant chemoradiotherapy

INTERVENTIONS:
Other: neoadjuvant chemoradiotherapy

SUMMARY:
For now, neoadjuvant chemoradiotherapy is routinely performed for T3N1-2M0 rectal cancer. However, there are lots of complications following neoadjuvant chemoradiotherapy, such as Wound-related complications, anastomotic leakage, anastomotic stenosis, sexual dysfunction, testicular or ovary failure. Patients undergoing resection for rectal cancer had low rates of local recurrence and long disease-free survival regardless of whether an APR, CAA or low AR was performed. The main purpose of preoperative radiotherapy is to lower the local recurrence. For the T3N1-2M0 rectal cancer with negative circumferential resection margin based on MRI assessment, we suppose might not necessary to receive neoadjuvant chemoradiotherapy, for operation can achieve the negative circumferential resection margin.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor within 12 cm of the anal verge
2. T3N1-2 as determined by preoperative MRI examination
3. negative circumferential resection margin determined by preoperative MRI examination
4. Absence of distant metastases
5. Absence of intestinal obstruction

Exclusion Criteria:

1. With distant metastases
2. With intestinal obstruction
3. Pregnancy or lactation
4. With operation contraindication
5. With mental disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
circumferential resection margin | one week after operation
introperative perforation | During the operation

SECONDARY OUTCOMES:
local recurrece | 3 years after operation
overal survival | 3 years after operation
disease-free survival | 3 years after operation
complications | 30 days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China